CLINICAL TRIAL: NCT04484753
Title: Validation of the iPelvis Mobile Application for Pelvic Physiotherapy in Women With Female Pelvic Floor Dysfunction
Brief Title: Validation of iPelvis App for Female Pelvic Floor Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rogério de Fraga (Other)
Responsible Party: Sponsor-Investigator, Rogério de Fraga, director, Faculdade Inspirar
Organization: Faculdade Inspirar (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Faculdade Inspirar
Record Dates: First submitted 2017-12-14; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Female Sexual Dysfunction; Urinary Incontinence
Keywords: urinary incontinence; female sexual dysfunction; quality of life; adherence; pelvic physiotherapy; post-partum
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- Home Exercise Sheet (Other): The participant took the sheet with the description of the exercises to his address.
  Interventions: Other: Home Exercise Sheet
- Ipelvis mobile application (Other): The participant received the app and performs home exercises guided by the app.
  Interventions: Other: Ipelvis mobile application
- Home exercise sheet + Pelvic Physiotherapy (Active Comparator): The participant did group physical therapy and used the exercise sheet at home on other days.
  Interventions: Behavioral: Home exercise sheet + Pelvic Physiotherapy
- Ipelvis mobile application + Pelvic Physiotherapy (Active Comparator): The participant did group physical therapy and used the mobile application on other days.
  Interventions: Behavioral: Ipelvis mobile application + Pelvic Physiotherapy

INTERVENTIONS:
Other: Home Exercise Sheet — Received a sheet with pelvic floor muscle training guidelines to be performed at home. After 3 months all volunteers were reevaluated.
  Arms: Home Exercise Sheet
Other: Ipelvis mobile application — Received the iPelvis® Application with pelvic floor muscle training guidelines to be performed at home. After 3 months all volunteers were reevaluated.
  Arms: Ipelvis mobile application
Behavioral: Home exercise sheet + Pelvic Physiotherapy — Performed 12 Pelvic Physiotherapy sessions, in group, once a week and received a sheet with pelvic floor muscle training guidelines to be performed at home. After 3 months all volunteers were reevaluated.
  Arms: Home exercise sheet + Pelvic Physiotherapy
Behavioral: Ipelvis mobile application + Pelvic Physiotherapy — Performed 12 pelvic physiotherapy sessions, in group, once a week and received the iPelvis® Application with pelvic floor muscle training guidelines to be performed at home. After 3 months all volunteers were reevaluated.
  Arms: Ipelvis mobile application + Pelvic Physiotherapy

SUMMARY:
The iPelvis app aims to improve adherence to pelvic physiotherapy on women with pelvic floor related dysfunctions, such as urinary or fecal incontinence, sexual dysfunction, etc.

DETAILED DESCRIPTION:
Urinary dysfunctions are widely discussed because they cause problems in social, emotional, sexual life and the quality of life of incontinent women. The overall objective of this research is to evaluate the use of the Application. Ipelvis in women with urinary incontinence. This is a longitudinal study of the type randomized controlled trial. Women with urinary incontinence of urgency, effort and effort will be evaluated and treated. Frequently asked questions, questions and answers, Quality of Life Questionnaires, Health Requirements, ICIQ-SF, ICIQ-OAB, FSFI and evaluation of pelvic, manual and electromyographic floor musculature function. As volunteers are drawn in four groups (Group I: Household Exercise Sheet / Group II: Ipelvis application / Group III: Household Exercise Sheet + Pelvic Physiotherapy / Group IV Ipelvis Application + Pelvic Physiotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Women with urinary incontinence by urodynamics, stress and mixed urinary incontinence, aged between 18 and 59 years, who have cognitive ability, have a compatible cell to install the Ipelvis application and who sign the Informed Consent Form.

Exclusion Criteria:

* Pregnant women, women up to six months postpartum, women with prolapse greater than stage III by Pelvic Organ Prolapse - Quantification (POP-Q), women with urinary tract infection, women with pelvic pain Performing therapies offered or having undergone pelvic surgery within a period of less than six months; With a pacemaker or contraceptive device (IUD); Women with intrapelvic tumor.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | 3 Months
  A tool that assesses the impact of UI on the quality of life and severity of urinary symptoms. The questionnaire is composed of four questions related to frequency, severity of urinary loss and its impact on quality of life. The ICIQ score is the sum of the scores from questions three, four and five and ranges from 0 to 21.

SECONDARY OUTCOMES:
Kings Health Questionnaire (KHQ) | 3 Months
  A questionnaire that analyzes the presence of Urinary Incontinence symptoms and their impact on various aspects of individuality in quality of life. The questionnaire is composed of 30 questions subdivided into nine domains. They report, respectively, the general perception of health, the impact of incontinence, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep and energy, and severity measures. To achieve the overall KHQ score, some pre-established calculations were performed, which provided scores for subsequent correlations.
The Female Sexual Function Index (FSFI) | 3 Months
  The questionnaire consists of 19 questions, which provide information on five domains of sexual response: desire and subjective stimulation, lubrication, orgasm, satisfaction and pain or discomfort. Individual scores are considered by the sum of items that comprise each domain (simple score), which are multiplied by the factor of that domain and can be explored or weighted. A final score (total scores: minimum of 2 and maximum of 36) is the total value of weighted scores for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Rogério Fraga, Study Director — Faculdade Inspirar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322